CLINICAL TRIAL: NCT03066115
Title: Contributions of Nitric Oxide Synthase, Cyclooxygenase, and Reactive Oxygen Species to Regional Cerebrovascular Control During Hypoxia and Hypercapnia
Brief Title: Impact of NOS, COX, and ROS Inhibition on Cerebral Blood Flow Regulation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was never funded, never fully IRB approved, and thus never enrolled anyone.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-1014
Record Dates: First submitted 2017-02-22; First posted 2017-02-28 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Hypoxia; Hypercapnia
Keywords: Cerebral blood flow; Cyclooxygenase; Nitric oxide synthase; Reactive Oxygen Species
MeSH Terms: conditions — Hypoxia; Hypercapnia | interventions — omega-N-Methylarginine; Ketorolac; Ascorbic Acid; Ultrasonography, Doppler, Transcranial; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NOS, COX, and ROS Inhibition (Experimental): Subjects will receive L-NMMA, ketorolac, then ascorbic acid via intravenous catheter. L-NMMA will have a 3 mg kg-1 loading dose over 5-minutes (36 mg kg-1 hr-1), followed by a maintenance dose of 1 mg kg-1 hr-1. Ketorolac will have a 0.3 mg kg-1 loading dose over 5 minutes (3.6 mg kg-1 hr-1) with a minimum loading dose of 15 mg. This will be followed by a maintenance dose of 0.03 mg kg-1 hr-1. Ascorbic acid will have a loading dose of 0.035 g kg fat-free mass-1 over 5-minutes (0.42 g kg fat-free mass-1 hr-1), followed by a maintenance dose of 0.060 g kg fat-free mass-1 hr-1. Cerebral blood flow velocity will be measured throughout the drug infusions via transcranial Doppler ultrasound.
  Interventions: Drug: L-NMMA; Drug: Ketorolac; Drug: Ascorbic Acid; Procedure: Intravenous Catheter; Procedure: Transcranial Doppler Ultrasound
- COX, NOS, and ROS Inhibition (Experimental): Subjects will receive ketorolac, L-NMMA, then ascorbic acid via intravenous catheter.
  Ketorolac will have a 0.3 mg kg-1 loading dose over 5 minutes (3.6 mg kg-1 hr-1) with a minimum loading dose of 15 mg. This will be followed by a maintenance dose of 0.03 mg kg-1 hr-1. L-NMMA will have a 3 mg kg-1 loading dose over 5-minutes (36 mg kg-1 hr-1), followed by a maintenance dose of 1 mg kg-1 hr-1. Ascorbic acid will have a loading dose of 0.035 g kg fat-free mass-1 over 5-minutes (0.42 g kg fat-free mass-1 hr-1), followed by a maintenance dose of 0.060 g kg fat-free mass-1 hr-1. Cerebral blood flow velocity will be measured throughout the drug infusions via transcranial Doppler ultrasound.
  Interventions: Drug: L-NMMA; Drug: Ketorolac; Drug: Ascorbic Acid; Procedure: Intravenous Catheter; Procedure: Transcranial Doppler Ultrasound

INTERVENTIONS:
Drug: L-NMMA — See arm description.
  Other Names: NOS Inhibition
Drug: Ketorolac — See arm description.
  Other Names: COX Inhibition
Drug: Ascorbic Acid — See arm description.
  Other Names: ROS Inhibition
Procedure: Intravenous Catheter — Two intravenous catheters will be placed for each study visit. One catheter will be used for the intravenous infusion of study drugs (L-NMMA, Ketorolac, and Ascorbic Acid). The second catheter will be used to draw intermittent blood samples at 8-specific time points throughout each study visit to ensure pharmaceutical efficacy and examine systemic physiologic blood variables of interest.
  Other Names: Cath
Procedure: Transcranial Doppler Ultrasound — MCAv will be measured via the transtemporal window while BAv will be measured through the transforaminal window with 2-MHz transcranial Doppler ultrasound probes (TCD, Neurovision model 500M, Multigon Industries, Inc.; Yonkers, NY, USA)
  Other Names: Ultrasound

SUMMARY:
Elucidating cerebrovascular control mechanisms during physiologic stress may help identify novel therapeutic targets aimed at preventing or reducing the impact of cerebrovascular disease. The physiological stressors of hypoxia and hypercapnia will be utilized to elicit increases in cerebral blood flow (CBF), and intravenously infused drugs will allow for the testing of potential mechanisms of cerebrovascular control. Specifically, the contributions of nitric oxide synthase (NOS), cyclooxygenase (COX), and reactive oxygen species (ROS) to hypoxic and hypercapnic increases in CBF will be examined. The concept that these mechanisms interact in a compensatory fashion to ensure adequate CBF during both hypoxia and hypercapnia will also be tested.

~25 young, healthy men and women will be tested at rest and during hypoxia and hypercapnia. Subjects will participate in two randomized, counterbalanced study visits under the following conditions: inhibition of NOS, NOS-COX, and NOS-COX-ROS or inhibition of COX, COX-NOS, COX-NOS-ROS. During hypoxia, arterial oxygen saturation will be lowered to 80% and end-tidal carbon dioxide will be maintained at basal levels. During hypercapnia arterial carbon dioxide will be increased ~10 mmHg above basal levels and arterial oxygen saturation will be maintained. Blood flow velocity will be measured with transcranial Doppler ultrasound in the anterior (middle cerebral artery; MCA) and posterior (basilar artery; BA) circulations as a surrogate for CBF.

It is hypothesized that both NOS and COX independently contribute to hypoxic and hypercapnic vasodilation in the MCA and BA, combined NOS-COX contribute to hypoxic and hypercapnic vasodilation in MCA and BA to a greater extent than either NOS or COX alone, and NOS-COX-ROS contribute to hypoxic and hypercapnic vasodilation in the MCA and BA to a greater extent than NOS-COX.

DETAILED DESCRIPTION:
Specific Aims:

1A. Determine the independent contributions of NOS and COX to hypoxic and hypercapnic vasodilation in the MCA of young, healthy adults.

1B. Determine the combined contribution of NOS and COX to hypoxic and hypercapnic vasodilation in the MCA of young, healthy adults.

1. C. Determine the combined contribution of NOS, COX, and ROS to hypoxic and hypercapnic vasodilation in the MCA of young, healthy adults.
2. A. Determine the independent contributions of NOS and COX to hypoxic and hypercapnic vasodilation in the BA of young, healthy adults.

2B. Determine the combined contribution of NOS and COX to hypoxic and hypercapnic vasodilation in the BA of young, healthy adults.

2C. Determine the combined contribution of NOS, COX, and ROS to hypoxic and hypercapnic vasodilation in the BA of young, healthy adults.

Initial Screening: A phone screening questionnaire will determine whether or not potential subjects meet preliminary eligibility criteria. Potentially eligible subjects will be invited for an additional in-person screening. Subjects will need to come to the screening visit having fasted (except water) for a minimum of 10 hours.

Laboratory screening procedures include:

1. Informed consent
2. Health history questionnaire
3. Physical activity questionnaire
4. Urine pregnancy test (females only)
5. Venous blood draw
6. DEXA scan (dual energy x-ray absorptiometry)

Study Design: Eligible subjects will complete 2 study visits examining hypoxic and hypercapnic responses under four conditions: control, NOS inhibition or COX inhibition, NOS and COX inhibition and NOS, COX, and ROS inhibition. During visit 1, subjects will receive L-NMMA (NG-Monomethyl-L-arginine; NOS inhibition), ketorolac (COX inhibition), then ascorbic acid (ROS inhibition). During visit 2, subjects will receive ketorolac, L-NMMA, then ascorbic acid. Study visits will be conducted in a randomized, counterbalanced order and all drugs will be infused intravenously. Hypoxia will elicit an SPO2~80% as determined by pulse oximetry and hypercapnia will increase end-tidal CO2 (PETCO2) by ~10 mmHg from baseline. Throughout each visit, subjects will be monitored for heart rate, blood pressure, pulse oximetry oxygen saturation, respiratory gases, ventilation, and CBF velocity. After instrumentation and baseline data collection, hypoxic and hypercapnic trials will commence with middle cerebral artery velocity (MCAv), basilar artery velocity (BAv), respiratory, and cardiovascular variables being recorded. All trials will be separated by 10-minutes of quiet rest while breathing room air and will not be randomized due to the order and timing of drug infusions required to explore our aims. Due to the difficulty of insonating the BA, this will serve as an exploratory aim and not deemed a necessary outcome for study completion.

Experimental Methods and Intervention Plan:

Transcranial Doppler Ultrasound (TCD) MCAv will be measured via the transtemporal window while BAv will be measured through the transforaminal window with 2-MHz (megahertz) transcranial Doppler ultrasound probes. In approximately 30% of individuals the BA cannot be identified; therefore, insonation of the MCA alone will be deemed sufficient to proceed with the study in cases in which BA cannot be located.

Measurements Height and weight will be measured to calculate body mass index (BMI). Waist and hip circumferences will be measured as indicators of regional adiposity. DEXA scan will be used for determination of body composition. Venous blood samples will be obtained for the determination of blood chemistry values. During each visit, subjects will be studied in a semi-recumbent position and instrumented for continuous measurement of heart rate (3-lead ECG), pulse oximetry oxygen saturation (SPO2, pulse oximeter), and blood pressure (MABP, automated physiological monitor). Hemodynamic parameters will be continuously measured with finger plethysmography. Inspiratory and expiratory gases will be measured with a gas analyzer and respiratory flow will be determined with a heated pneumotachometer.

Hypoxia Hypoxia will be used to cause cerebral vasodilation under resting, semi-recumbent conditions. Three isocapnic hypoxia trials will be performed per study visit. Subjects will inspire through a two-way non-rebreathing valve, connected to a gas mixer, supplied by medical grade pressurized oxygen (O2), carbon dioxide (CO2), and nitrogen (N2). After 3-minutes of baseline room air breathing, hypoxia will be introduced by decreasing inspired O2 (~11% O2) to elicit and sustain 3-minutes of SPO2~80% as determined by a pulse oximeter. After 3-minutes of baseline steady state hypoxia, there will be a 5-minute drug loading period (L-NMMA, ketoroloc, or ascorbic acid), followed by a 5-minute drug maintenance period. Hypoxia will be maintained during this time, with total hypoxia duration of ~15-minutes per each hypoxia trial. Isocapnia will be achieved through the addition of CO2 to inspired gas. End-tidal CO2 (PETCO2) has been shown to be a valid predictor of arterial blood CO2 levels. Prior data from our lab indicate that steady state hypoxia is achieved within 3 minutes. Additionally, hypoxia eliciting an SPO2~80% will be examined as cerebral vessels have relatively low cerebrovascular sensitivity to less severe hypoxia (SPO2~90%). A total of 3 hypoxia trials will be conducted per study visit yielding ~45 minutes of steady state hypoxia.

Hypercapnia An increase in systemic CO2 is a powerful signal to increase blood flow within the cerebral circulation. A total of 4 hypercapnic trials will be performed during each study visit. Subjects will inspire through a three-way sliding rebreathing valve attached to a latex balloon containing a hyperoxic (O2=40%), hypercapnic (CO2=3%) gas mixture with the balance N2. The balloon will be filled to a volume exceeding estimated vital capacity (as determined by age, sex, and height) by 1-liter. After 3-minutes of baseline room air breathing, hypercapnia will commence by sliding the three-way rebreathing valve from room air to the attached latex balloon. During hypercapnia, PETCO2 increases (~10 mmHg above baseline values), but inspired O2 does not fall below room air percentage of 21%. Hypercapnia will be sustained (~2-minutes) until PETCO2 values reach ~10 mmHg above baseline values, after which subject will begin breathing room air. PETCO2 will be used as a reliable, non-invasive measure of arterial CO2. A total of 4 hypercapnic trials will be conducted per study visit yielding ~ 8 minutes of hypercapnia per study visit.

Intravenous Catheter Trained lab personnel will place two intravenous catheters (one in each arm) for each study visit. One catheter will be used for the intravenous infusion of study drugs (L-NMMA, Ketorolac, and Ascorbic Acid). The second catheter will be used to draw intermittent blood samples at 8-specific time points throughout each study visit to ensure pharmaceutical efficacy and examine systemic physiologic blood variables of interest. The catheter used for blood draws will be kept patent with a 0.9% saline drip. If only one IV catheter can be placed or one fails, the study will proceed with both drug infusion and blood draws occurring from a single catheter.

Intravenous L-NMMA Infusion Intravenous L-NMMA is the only non-FDA approved drug that will be used, but is commonly utilized in the research setting. Intravenous infusion of L-NMMA will be used to inhibit the enzyme NOS which is responsible for the formation of NO. L-NMMA is a lyophilized powder that is diluted with saline. In the current study, intravenous L-NMMA will be administered via a 3 mg kg-1 loading dose over 5-minutes (36 mg kg-1 hr-1), followed by a maintenance dose of 1 mg kg-1 hr-1 for the remainder of the study. Considering a typical 75 kg individual this will result in a loading dose of 225mg and a maintenance dose (~112min) of 140mg totaling 365 mg L-NMMA throughout the duration of the study, when L-NMMA is the first study drug infused (L-NMMA infused during HX1, HX2, HX3 and HC2, HC3, HC4). During the visit when L-NMMA is second study drug infused (L-NMMA infused during HX2, HX3 and HC3, HC4) the total dosing will be less as the maintenance infusion (~67 min) will be reduced by ~45 minutes totaling 309 mg L-NMMA. The loading dose of L-NMMA is equivalent to that used in a prior study investigating the contribution of NOS to hypoxic cerebral vasodilation while the maintenance dose and the absolute amount of L-NMMA infused will be less than previously utilized.

Intravenous Ketorolac Infusion Intravenous ketorolac is FDA approved non-steroidal anti-inflammatory drug used for the treatment of pain. Ketorolac will be used to non-specifically inhibit the enzyme cyclooxygenase which is responsible for the formation of vasoactive prostaglandins (prostacyclin, thromboxane). Inhibition of prostaglandin synthesis during hypoxia will allow assessment of the contribution of these vasoactive prostaglandins to hypoxic vasodilation. Common intravenous doses of ketorolac are 15 mg and 30 mg bolus infusions; however, ketorolac will be dosed relative to body mass. Ketorolac will be intravenously administered via a 0.3 mg kg-1 loading dose over 5 minutes (3.6 mg kg-1 hr-1) with a minimum loading dose of 15 mg. This will then be followed by a maintenance dose of 0.03 mg kg-1 hr-1 for the remainder of the study. Considering a typical 75 kg individual this will result in a loading dose of 22.5 mg and a maintenance dose (~112min) of 4.2 mg totaling 26.7 mg ketorolac throughout the duration of the study, when ketorolac is the first study drug infused (ketorolac infused during HX1, HX2, HX3 and HC2, HC3, HC4). During the visit when ketorolac is second study drug infused ketorolac infused during HX2, HX3 and HC3, HC4) the total dosing will be less as the maintenance infusion (~67 min) will be reduced by ~45 minutes totaling 25 mg of ketorolac. Similar doses of ketorolac have been shown to reduce whole body prostanoids and reduce perioperative pain. Plasma ketorolac concentrations peak within ~3 minutes following intravenous administration with a terminal half-life of 5.6 hours.

Intravenous Ascorbic Acid Infusion Intravenous ascorbic acid is FDA-approved. Ascorbic acid will be intravenously administered to acutely reduce ROS. Ascorbic acid will be administered via loading dose of 0.035 g kg fat-free mass-1 over 5-minutes (0.42 g kg fat-free mass-1 hr-1). Followed by a maintenance dose of 0.060 g kg fat-free mass-1 hr-1 over the remaining study time course (~20 minutes) for continued suppression of reactive oxygen species. Considering a 75 kg individual with a fat-free tissue mass of ~55kg (based upon previous young, healthy subjects in our lab), subjects will receive ~ 3.025 g of Ascorbic acid during the course of a study visit.

Plasma Assays

~10 mL of blood will be drawn during the screening visit as a component of study eligibility. Screening blood samples will be analyzed for fasting venous glucose, creatinine, total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides. Venous blood samples will be drawn at 8 time points during the study protocol via a venous catheter. Each blood draw will be 10 mL, totaling 80 mL. Blood will be centrifuged with plasma and serum drawn off and stored at -80ºC. Efficacy of COX inhibition will be determined by the measurement (EIA) of the circulating COX metabolites 6-keto-prostaglandin F1α (as stable marker of PGI2) and thromboxane B2 (a stable marker of TXA2). Efficacy of ROS inhibition will be determined by plasma vitamin C concentrations and oxidized low-density lipoproteins (oxLDL) serving as a systemic marker of oxidative stress. Acute intravenous Ascorbic acid administration has been shown to decrease oxLDL in healthy adults. Efficacy of NOS inhibition will be determined by sum of nitrite and nitrate (NOx), which is considered to be an index of NO production.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 ≤ years ≤ 45
2. Free of disease and otherwise healthy as determined by health history questionnaire
3. Not currently taking medication with the exception of birth control as determined by health history questionnaire
4. Low to moderate physical activity will be permitted and assessed by a physical activity questionnaire (≤ 4 hours of physical activity/week)
5. Body mass index (BMI) < 25 kg/m2
6. Resting blood pressure <140/<90 mmHg (lowest of three measures)
7. Resting heart rate <100 bpm
8. Resting pulse oximetry oxygen saturation (SPO2) >95%
9. Fasting venous blood values (average of two measures)

   1. Glucose <100 mg/dL
   2. Creatinine < 1.5 mg/dL
   3. Total cholesterol <200 mg/dL

   i. HDL cholesterol >40 mg/dL (men) ii. HDL cholesterol >50 mg/dL (women) iii. LDL cholesterol < 130 mg/dL d. Triglycerides <150 mg/dL
10. Subjects must be willing to report to the laboratory on all study days after completing

    1. Minimum 10-hour fast
    2. Minimum 18-hours abstention from exercise, alcohol, caffeine, and non-steroidal anti-inflammatory drugs (i.e. aspirin, ibuprofen, and naproxen)
11. Additionally, women will

    1. Have a regular menstrual cycle (self-report)
    2. Be studied (study visit 1 and study visit 2) on days 1-5 of menstrual cycle (self- report).

Exclusion Criteria:

1. Coronary artery disease
2. Stroke
3. Heart attack
4. Heart valve disease
5. Congestive heart failure
6. Previous heart surgery
7. Lung disease
8. Peripheral vascular disease
9. Gastrointestinal (GI) bleeding
10. Allergy or Intolerance to Aspirin or NSAIDS
11. History of renal/kidney disease, insufficiency, or injury
12. Smoke or use tobacco within the last year
13. Subject has an abnormality or contraindication to study participation, which is not covered in the eligibility criteria.

Additionally, women will be excluded if they are

1. Pregnant (as determined by a urine pregnancy test on screening and study days)
2. Currently breastfeeding (self-report)
3. Post-menopausal (self-report)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral blood flow velocity in the middle cerebral artery | Through study completion (up to 1 year)
  How cerebral blood flow velocity changes during hypoxia or hypercapnia with COX, NOS, and ROS inhibition in the middle cerebral artery as measured by transcranial Doppler ultrasound.

SECONDARY OUTCOMES:
Change in cerebral blood flow velocity in the basilar artery | Through study completion (up to 1 year)
  How cerebral blood flow velocity changes during hypoxia or hypercapnia with COX, NOS, and ROS inhibition in the basilar artery as measured by transcranial Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: William G Schrage, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No